CLINICAL TRIAL: NCT03448887
Title: Cardiovascular Risk Comparison Between Expanded Hemodialysis Using Theranova and On-line Hemodiafiltration - Exploratory, Multicenter, Randomized Clinical Trial
Brief Title: Cardiovascular Risk Comparison Between Expanded Hemodialysis Using Theranova and On-line Hemodiafiltration
Acronym: CARTOON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Seoul St. Mary's Hospital (Other); Seoul National University Bundang Hospital (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Kwon wook Joo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Theranova-SNU-01
Record Dates: First submitted 2018-02-16; First posted 2018-02-28 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Kidney Failure, Chronic; Renal Dialysis
Keywords: End-stage renal disease; Medium cut-off dialyzer; Hemodiafiltration; Cardiovascular; Pulse wave velocity
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Exploratory, Multicenter, Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study group (Experimental): Extended HD with MCO dialyzer
  Interventions: Device: Theranova
- Control group (Active Comparator): Online hemodiafiltration
  Interventions: Device: Online hemodiafiltration

INTERVENTIONS:
Device: Theranova — Extended HD with theranova
  Arms: Study group
Device: Online hemodiafiltration — Online hemodiafiltration
  Arms: Control group

SUMMARY:
Theranova is a novel medium cut-off (MCO) dialyzer. Previous studies identified that theranova dialyzer had superior performance on middle molecule removal to conventional hemodialysis (HD) and hemodiafiltration (HDF). The present study addresses to compare clinical outcomes including cardiovascular endpoint between HD with theranova dialyzer and HDF.

DETAILED DESCRIPTION:
While conventional hemodialysis (HD) modality effectively removes small-sized molecules, performance with middle-sized and protein-bound molecules is not well established. With increasing perception on importance of middle molecule removal, on-line hemodiafiltration (HDF) is getting more attention from healthcare professionals. However, HDF has not been widely used in Korea due to its technical burden and limited public funding issue.

Novel medium cut-off (MCO) dialyzer, Theranova, is available in Korea, which showed superior performance on middle molecule removal to conventional HD and HDF from the previous study. This new dialyzer can be a good alternative option replacing conventional HD or even HDF with its benefits. However, current data available on the MCP dialyzer has certain limitations such as small sample size, no Asian subject included, limited types of biomarkers, and no clinical outcomes (particularly cardiovascular diseases) included.

With this respect, performance comparison of MCO dialyzer with HDF in terms of clinical outcomes, including cardiovascular endpoint would fill the exiting data gap, which is absolutely important to make a clinical decision on dialysis modality.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Hemodialysis more than 3 months because of end-stage renal disease
* Consent to the study protocol

Exclusion Criteria:

* Already receiving online hemodiafiltration before study enrollment
* Dialysis schedule other than three times per week (e.g., once per week)
* Receiving concurrent peritoneal dialysis
* Having a plan to receive kidney transplantation within 1 year
* Having multiple myeloma or monoclonal gammopathy
* Having advanced or active malignancy
* Having a plan to be pregnant or being pregnant / breast-feeding or not having a plan to use contraception
* Participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in cardiovascular surrogate marker | 0, 6, 12 months
  Brachial-ankle pulse wave velocity (m/s)

SECONDARY OUTCOMES:
Change in cardiac surrogate marker #1 | 0, 6, 12 months
  CT coronary calcium scoring (score)
Change in cardiac surrogate marker #2 | 0, 6, 12 months
  Echocardiography: ejection fraction (%); E/e' ratio (cm/s per cm/s); LVMI (g/m2).
Change in cardiovascular biomarkers #1 | 0, 6, 12 months
  Plasma levels of BNP (pg/ml)
Change in cardiovascular biomarkers #2 | 0, 6, 12 months
  Plasma levels of NT-proBNP (pg/ml)
Change in cardiovascular biomarkers #3 | 0, 6, 12 months
  Plasma levels of hsCRP (mg/dl)
Change in cardiovascular biomarkers #4 | 0, 6, 12 months
  Plasma levels of troponin-I (ng/ml)
Change in cardiovascular biomarkers #5 | 0, 6, 12 months
  Plasma levels of troponin-T (ng/ml)
Change in cardiovascular biomarkers #6 | 0, 6, 12 months
  Plasma levels of IL-6 (pg/ml)
Patient-reported outcomes #1 | 0, 6, 12 months
  Dialysis symptom index (score)
Patient-reported outcomes #2 | 0, 6, 12 months
  Degree of fatigue after dialysis (scale from 0 to 10)
Patient-reported outcomes #3 | 0, 6, 12 months
  Post-dialysis recovery time (within minutes, when arriving home, at bed time, next morning, by next dialysis)

CONTACTS AND LOCATIONS:
Overall Officials: Kwon Wook Joo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kirsch AH, Lyko R, Nilsson LG, Beck W, Amdahl M, Lechner P, Schneider A, Wanner C, Rosenkranz AR, Krieter DH. Performance of hemodialysis with novel medium cut-off dialyzers. Nephrol Dial Transplant. 2017 Jan 1;32(1):165-172. doi: 10.1093/ndt/gfw310. PMID 27587605